CLINICAL TRIAL: NCT00480896
Title: Clinical Study on Tacrolimus Ointment Over the Long-term. "CONTROL Study - Children"
Brief Title: Treatment and Control of Atopic Dermatitis With 0.03% Tacrolimus Ointment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FG-506-06-41
Record Dates: First submitted 2007-05-30; First posted 2007-05-31 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Dermatitis, Atopic
Keywords: Dermatitis, atopic; Tacrolimus; Child; treatment outcomes
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Tacrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: tacrolimus ointment
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo ointment

INTERVENTIONS:
Drug: tacrolimus ointment — Topical application
  Other Names: Protopic®; FK506 ointment
  Arms: 1
Drug: Placebo ointment — Topical application
  Arms: 2

SUMMARY:
A long-term 0.03% tacrolimus ointment based regimen comprising of up to 6 weeks of initial twice daily treatment and subsequent twice weekly prophylactic application can effectively treat active lesions of atopic dermatitis, and prevent, delay, and reduce flares.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient of any ethnic group
* Patient was at least 2-15 years old and suffered from mild to severe atopic dermatitis (Rajka/Langeland score of at least 3)

Exclusion Criteria:

* Patient had a genetic epidermal barrier defect such as Netherton's syndrome or generalised erythroderma
* Patient had a clinically significant skin infection on the affected (and to be treated) area

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Actual)
Dates: Start 2004-06; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Number of exacerbations of atopic dermatitis requiring intervention. | 12 months

SECONDARY OUTCOMES:
Time to first exacerbation requiring intervention; exacerbation treatment days, periods and time to first exacerbation; physician and patient assessment of affected area, treatment response; quality of life; global response. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Principal Investigator — Universitätsklinikum Frankfurt Zentrum für Dermatologie
Locations (22):
- Brussels, Belgium
- Czechia (2):
  - Brno
  - 3 Sites, Prague
- Helsinki, Finland
- France (2):
  - Nantes
  - Paris
- Germany (4):
  - Düsseldorf
  - Frankfurt
  - Kiel
  - Mahlow
- Budapest, Hungary
- Italy (3):
  - Bergamo
  - Parma
  - Roma
- Netherlands (4):
  - Amsterdam
  - Groningen
  - Nijmegen
  - Utrecht
- Porto, Portugal
- Barcelona, Spain
- United Kingdom (2):
  - Birmingham
  - London

REFERENCES:
- [Background] Thaci D, Reitamo S, Gonzalez Ensenat MA, Moss C, Boccaletti V, Cainelli T, van der Valk P, Buckova H, Sebastian M, Schuttelaar ML, Ruzicka T; European Tacrolimus Ointment Study Group. Proactive disease management with 0.03% tacrolimus ointment for children with atopic dermatitis: results of a randomized, multicentre, comparative study. Br J Dermatol. 2008 Dec;159(6):1348-56. doi: 10.1111/j.1365-2133.2008.08813.x. Epub 2008 Sep 6. PMID 18782319